CLINICAL TRIAL: NCT02444039
Title: Slit Lamp Model SL-D-301 and DC-4 Digital Camera Attachment
Brief Title: Slit Lamp and Digital Camera Attachment
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: TOPCON-004-2014
Record Dates: First submitted 2014-11-20; First posted 2015-05-14 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Any Willing and Able Person for Ocular Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Any Willing and Able Person for Ocular Imaging: Any Willing and Able Person for Ocular Imaging
  Interventions: Device: SL-D301; Device: DC-4; Device: SL-3G

INTERVENTIONS:
Device: SL-D301 — Slit Lamp
Device: DC-4 — Digital Camera Attachment
Device: SL-3G — Slit Lamp

SUMMARY:
The objective of the study is to compare the ease of use and performance of the SL-D301 with the DC-4 with other existing slit lamps imaging systems (SL-3G) from Topcon.

DETAILED DESCRIPTION:
The objective of the study is to compare the ease of use and performance of the SL-D301 with the DC-4 with other existing slit lamps imaging systems (SL-3G) from Topcon and ascertain that the changes and new features incorporated do not interfere with the normal use and application of the device.

ELIGIBILITY:
Inclusion Criteria:

* Any willing subject

Exclusion Criteria:

* Subjects unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any Willing and able subjects will be recruited from Topcon Medical Systems.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Instrument and Device Evaluation | 1 Hour

CONTACTS AND LOCATIONS:
Overall Officials: Danny Leung, Principal Investigator — Topcon Corporation
Locations (1):
- Topcon Medical Systems, Inc., Oakland, New Jersey, United States